CLINICAL TRIAL: NCT01296711
Title: A Phase 2, Multicenter, Open-Label, Follow-up Study to Assess the Long-Term Safety and Efficacy of CDP6038 (Olokizumab) Administered Subcutaneously to Subjects With Active Rheumatoid Arthritis Who Completed Study RA0056
Brief Title: Open-label Study to Assess the Safety and Efficacy of CDP6038 (Olokizumab) in Patients Who Completed RA0056
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Decision to out-license the compound for further development
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Collaborators: R-Pharm (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RA0057; 2010-022224-77 (EudraCT Number)
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Results first posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; CDP6038; Interleukin-6
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — olokizumab

STUDY DESIGN:
Intervention Model Description: RA0057 is a single arm study, however, analyses will also be performed according to the original treatment arms of the parent study RA0056 (NCT01242488).
Oversight: Data Monitoring Committee: No

ARMS (1):
- CDP6038 (olokizumab) (Experimental)
  Interventions: Biological: CDP6038 (olokizumab)

INTERVENTIONS:
Biological: CDP6038 (olokizumab) — 100mg/ml solution for injection 120 mg subcutaneously (sc) every 2 weeks

SUMMARY:
The purpose of this study is to evaluate the long term safety and tolerability of CDP6038 (olokizumab) treatment in adult subjects with active rheumatoid arthritis who completed study RA0056 (NCT01242488).

DETAILED DESCRIPTION:
Male and female subjects were randomized in a multi-center, open-label, follow-up study to assess the long-term safety and efficacy of a subcutaneous dose of 120 mg CDP6038 (olokizumab), every two weeks, for the treatment of active rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Subject completed the RA0056 study (Week 12 Visit)
* Subject must have maintained their stable dose (and route) of methotrexate (MTX) between 12.5 to 25mg/week in RA0056, and plan to maintain this same dose and route of administration for at least 12 weeks
* Female subjects must be either postmenopausal for at least 1 year, surgically incapable of childbearing, or effectively practicing an acceptable method of contraception (either oral/parenteral/implantable hormonal contraceptives, intrauterine device, or barrier and spermicide). Abstinence is not considered an acceptable method of contraception for this study
* Female subjects of childbearing potential must agree to use 2 methods of adequate contraception during the study and for 6 months (24 weeks) after their last CDP6038 (olokizumab) dose
* Male subjects must agree to ensure that they or their female partner(s) use adequate contraception during the study and for 12 weeks after the subject receives their last dose of CDP6038 (olokizumab)

Exclusion Criteria:

* Subject has an ongoing serious adverse event from the RA0056 study
* Female subject of childbearing potential has a positive pregnancy test at Week 12 in Study RA0056 or plans to become pregnant during the study or within 6 months (24 weeks) following their last dose of study medication
* Subject has evidence of active or latent tuberculosis
* Subject is receiving any biologic response modifier or synthetic disease-modifying antirheumatic drug other than MTX
* Subject has an alcohol consumption of more than 1 unit per weekday. One unit equals 1 glass of beer or lager (~330mL), a glass of wine (125mL), or a measure of spirits/hard liquor (25mL)
* Subject with any other condition in RA0056 (eg, clinically significant laboratory values, frequent adverse events) which in the Investigator's or Sponsor's judgment would make the subject unsuitable for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2011-03-07 (Actual); Primary Completion 2013-05-01 (Actual); Study Completion 2013-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Genovese, Dr, Principal Investigator — Stanford University
Locations (55):
- United States (50):
  - 166, Mesa, Arizona
  - 154, Phoenix, Arizona
  - 118, Scottsdale, Arizona
  - 103, Hot Springs, Arkansas
  - 127, Covina, California
  - 148, La Jolla, California
  - 184, Long Beach, California
  - 177, Los Angeles, California
  - 104, Palo Alto, California
  - 129, Santa Maria, California
  - 164, Upland, California
  - 141, Hamden, Connecticut
  - 111, Lewes, Delaware
  - 151, DeBary, Florida
  - 114, Jupiter, Florida
  - 157, Tampa, Florida
  - 183, Tampa, Florida
  - 116, Idaho Falls, Idaho
  - 160, Moline, Illinois
  - 168, Springfield, Illinois
  - 133, Cedar Rapids, Iowa
  - 172, Kansas City, Kansas
  - 185, Saint Clair Shores, Michigan
  - 112, St Louis, Missouri
  - 134, St Louis, Missouri
  - 102, Lincoln, Nebraska
  - 171, Freehold, New Jersey
  - 152, Toms River, New Jersey
  - 174, Brooklyn, New York
  - 170, Charlotte, North Carolina
  - 150, Cincinnati, Ohio
  - 100, Dayton, Ohio
  - 110, Oklahoma City, Oklahoma
  - 165, Duncansville, Pennsylvania
  - 105, Nashville, Tennessee
  - 135, Austin, Texas
  - 128, Dallas, Texas
  - 126, Houston, Texas
  - 132, Houston, Texas
  - 138, Houston, Texas
  - 181, Houston, Texas
  - 145, Mesquite, Texas
  - 143, Nassau Bay, Texas
  - 122, San Antonio, Texas
  - 144, Tomball, Texas
  - 142, Victoria, Texas
  - 139, Chesapeake, Virginia
  - 175, Tacoma, Washington
  - 136, Beckley, West Virginia
  - 167, Clarksburg, West Virginia
- Belgium (2):
  - 401, Brussels
  - 400, Liège
- United Kingdom (3):
  - 206, Essex
  - 208, Southampton
  - 209, Torquay

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The present study was an open-label extension to study RA0056 (NCT01242488). Subjects completing the 12-week treatment period of study RA0056 had the opportunity to participate in this study. First subject enrolled: 07 March 2011. Early termination: 05 Aug 2013.
Pre-assignment Details: 198 subjects completed the parent study RA0056 (NCT01242488); 190 subjects were enrolled in study RA0057. The study was a single treatment study and all subjects received CDP6038 (olokizumab) 120 mg sc q2w, however, some results are also presented according to the previously assigned treatment arms of the parent study RA0056.
Groups:
- RA0056 CDP6038 (Olokizumab) 120 mg q2w: CDP6038 (olokizumab) 120 mg administered every 2 weeks (q2w) sc in Study RA0056, and maintained at same dose (i.e. 120 mg q2w sc) at start of study RA0057 (Week 12 of RA0056) for 48 weeks.
- RA0056 CDP6038 (Olokizumab) 120 mg q4w: CDP6038 (olokizumab) 120 mg administered every 4 weeks (q4w) sc in Study RA0056, followed by switch to CDP6038 (olokizumab) 120 mg q2w sc at start of Study RA0057 (Week 12 of RA0056) for 48 weeks.
- RA0056 CDP6038 (Olokizumab) 240 mg q2w: CDP6038 (olokizumab) 240 mg administered q2w sc in study RA0056, followed by switch to CDP6038 (olokizumab) 120 mg q2w sc at start of Study RA0057 (Week 12 of RA0056) for 48 weeks.
- RA0056 CDP6038 (Olokizumab) 240 mg q4w: CDP6038 (olokizumab) 240 mg administered q4w sc in Study RA0056, followed by switch to CDP6038 (olokizumab) 120 mg q2w sc at start of Study RA0057 (Week 12 of RA0056) for 48 weeks.
- RA0056 CDP6038 (Olokizumab) 60 mg q2w: CDP6038 (olokizumab) 60 mg administered q2w sc in Study RA0056, followed by switch to CDP6038 (olokizumab) 120 mg q2w sc at start of Study RA0057 (Week 12 of RA0056) for 48 weeks.
- RA0056 CDP6038 (Olokizumab) 60 mg q4w: CDP6038 (olokizumab) 60 mg administered q4w sc in Study RA0056, followed by switch to CDP6038 (olokizumab) 120 mg q2w sc at start of Study RA0057 (Week 12 of RA0056) for 48 weeks.
- RA0056 Placebo: Placebo (sodium chloride, 0.9%) was administered q2w or q4w sc in Study RA0056, followed by switch to CDP6038 (olokizumab) 120 mg q2w sc at start of Study RA0057 (Week 12 of RA0056) for 48 weeks.
- RA0056 Tocilizumab 8 mg/kg q4w: Tocilizumab 8 mg/kg administered q4w iv in Study RA0056, followed by switch to CDP6038 (olokizumab) 120 mg q2w sc at start of Study RA0057 (Week 12 of RA0056) for 48 weeks.
Period: Overall Study
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Started | 20 | 20 | 21 | 20 | 17 | 16 | 40 | 36
Completed | 4 | 12 | 8 | 7 | 7 | 5 | 9 | 15
Not Completed | 16 | 8 | 13 | 13 | 10 | 11 | 31 | 21
Not completed — Adverse Event | 3 | 1 | 4 | 3 | 1 | 6 | 11 | 3
Not completed — Lack of Efficacy | 1 | 4 | 1 | 1 | 1 | 0 | 2 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 2 | 0 | 4 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 2 | 2 | 1 | 1 | 1 | 2 | 1
Not completed — Study termination | 8 | 1 | 5 | 4 | 4 | 4 | 8 | 10
Not completed — Continued elevated liver enzymes | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Methotrexate discontinued | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Investigator discretion | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Required restricted steroid injections | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Ongoing missed appointments | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Failure to comply with visits | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Patient decision due to transport | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population included all enrolled subjects who received at least 1 injection of CDP6038 (olokizumab) in Study RA0057.
Groups:
- RA0056 CDP6038 (Olokizumab) 120 mg q2w: CDP6038 (olokizumab) 120 mg administered q2w sc in Study RA0056, and maintained at same dose (i.e. 120 mg q2w sc) at start of Study RA0057 (Week 12 of RA0056) for 48 weeks.
- RA0056 CDP6038 (Olokizumab) 120 mg q4w: CDP6038 (olokizumab) 120 mg administered q4w sc in Study RA0056, followed by switch to CDP6038 (olokizumab) 120 mg q2w sc at start of Study RA0057 (Week 12 of RA0056) for 48 weeks.
- Total: Total of all reporting groups
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w | Total
Number analyzed (Participants) | 20 | 20 | 21 | 20 | 17 | 16 | 40 | 36 | 190
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 16 | 17 | 14 | 13 | 14 | 27 | 29 | 147
  >=65 years | 3 | 4 | 4 | 6 | 4 | 2 | 13 | 7 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 19 | 16 | 14 | 14 | 33 | 31 | 161
  Male | 3 | 3 | 2 | 4 | 3 | 2 | 7 | 5 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 3 | 2 | 1 | 4 | 3 | 4 | 19
  White | 19 | 18 | 18 | 18 | 16 | 12 | 35 | 31 | 167
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-emergent Adverse Events (TEAEs)
Description: Reported TEAEs included adverse events that started or worsened after the first dose of CDP6038 (olokizumab) in Study RA0057 and within 30 days after the last dose.
Time Frame: From Baseline (Week 0 of Study RA0057) until 30 days after the last dose (maximum up to 780 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 20 | 20 | 21 | 20 | 17 | 16 | 40 | 36
Participants | 17 | 20 | 19 | 18 | 15 | 15 | 39 | 35

2. Secondary Outcome: Change From Baseline (Week 0 of Study RA0056) in the Disease Activity Score-28-joint Count (C-reactive Protein) (DAS28[CRP]) to Week 12 of Study RA0057
Description: DAS28(CRP) was calculated using the tender/painful joint count (TJC) and swollen joint count (SJC) from 28 joints, the Patient's Global Assessment of Disease Activity (PtGADA)-Visual Analog Scale (VAS), andCRP according to the formula: DAS28(CRP)=0.56 * (TJC)^1/2 + 0.28 * (SJC)^1/2 + 0.36 * ln(CRP[mg/L]+1) + 0.014 * PtGADA + 0.96 Assessments: • TJC and SJC: assessed on the same 2-point scale (0=absent; 1=present). • PtGADA: 100 mm VAS (0=very good, no symptoms; 100=very poor, severe symptoms). • CRP value calculated in mg/L. The 28 joints included the shoulders, elbows, wrists; metacarpophalangeal (MCP), thumb interphalangeal (IP), and proximal interphalangeal (PIP) joints of the hands; and the knees. Scores on the DAS28(CRP) range from 0 to approximately 10, where higher scores indicate more disease activity. A negative change in DAS28(CRP) score indicates an improvement in disease activity.
Time Frame: Baseline (Week 0 of Study RA0056) and Week 12 (Study RA0057)
Population: Full Analysis Set (FAS) included all enrolled subjects who received at least 1 injection of CDP6038 (olokizumab) and in addition had at least 1 efficacy measurement in Study RA0057. When baseline and actual mean scores were not available, change from baseline was not calculated. Here, Number of Participants Analyzed included those participants who were evaluable for the assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 13 | 17 | 19 | 15 | 15 | 15 | 32 | 29
units on a scale | -2.2809 (1.45737) [lower limit 1.45737] | -2.2485 (1.39384) [lower limit 1.39384] | -2.5123 (1.39667) [lower limit 1.39667] | -2.2230 (1.17572) [lower limit 1.17572] | -1.6957 (0.67335) [lower limit 0.67335] | -2.1735 (1.56606) [lower limit 1.56606] | -2.3727 (1.41421) [lower limit 1.41421] | -2.4710 (1.43947) [lower limit 1.43947]

3. Secondary Outcome: Change From Baseline (Week 0 of Study RA0056) in DAS28(CRP) to Week 24 of Study RA0057
Description: DAS28(CRP) was calculated using the TJC and SJC from 28 joints, the PtGADA-VAS, and CRP according to the formula: DAS28(CRP)=0.56 * (TJC)^1/2 + 0.28 * (SJC)^1/2 + 0.36 * ln(CRP[mg/L]+1) + 0.014 * PtGADA + 0.96 Assessments: • TJC and SJC: assessed on the same 2-point scale (0=absent; 1=present). • PtGADA: 100 mm VAS (0=very good, no symptoms; 100=very poor, severe symptoms). • CRP value calculated in mg/L. The 28 joints included the shoulders, elbows, wrists; metacarpophalangeal (MCP), thumb interphalangeal (IP), and proximal interphalangeal (PIP) joints of the hands; and the knees. Scores on the DAS28(CRP) range from 0 to approximately 10, where higher scores indicate more disease activity. A negative change in DAS28(CRP) score indicates an improvement in disease activity.
Time Frame: Baseline (Week 0 of Study RA0056) and Week 24 (Study RA0057)
Population: FAS included all enrolled subjects who received at least 1 injection of CDP6038 (olokizumab) and in addition had at least 1 efficacy measurement in Study RA0057. When baseline and actual mean scores were not available, change from baseline was not calculated. Here, Number of Participants Analyzed included those participants who were evaluable for the assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 13 | 14 | 19 | 10 | 13 | 14 | 31 | 29
units on a scale | -2.6441 (1.46566) [lower limit 1.46566] | 1.46566 (1.17637) [lower limit 1.17637] | -2.5811 (1.40191) [lower limit 1.40191] | -2.5999 (1.16812) [lower limit 1.16812] | -1.7189 (0.87218) [lower limit 0.87218] | -2.4221 (1.37341) [lower limit 1.37341] | -2.1484 (1.34676) [lower limit 1.34676] | -2.7624 (1.47841) [lower limit 1.47841]

4. Secondary Outcome: Change From Baseline (Week 0 of Study RA0056) in DAS28(CRP) to Week 48 of Study RA0057
Description: as for outcome 3
Time Frame: Baseline (Week 0 of Study RA0056) and Week 48 (Study RA0057)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 10 | 12 | 13 | 10 | 12 | 10 | 20 | 22
units on a scale | -2.3257 (1.07427) [lower limit 1.07427] | -2.2498 (1.66580) [lower limit 1.66580] | -2.5277 (1.56763) [lower limit 1.56763] | -2.7050 (0.96160) [lower limit 0.96160] | -2.3824 (0.79065) [lower limit 0.79065] | -2.1501 (0.64141) [lower limit 0.64141] | -2.2403 (1.47765) [lower limit 1.47765] | -2.7611 (1.31329) [lower limit 1.31329]

5. Secondary Outcome: Change From Baseline (Week 0 of Study RA0056) in DAS28(CRP) to Week 96 of Study RA0057
Description: DAS28(CRP) was calculated using the TJC and SJC from 28 joints, the PtGADA-VAS, and CRP according to the formula: DAS28(CRP)=0.56 * (TJC)^1/2 + 0.28 * (SJC)^1/2 + 0.36 * ln(CRP[mg/L]+1) + 0.014 * PtGADA + 0.96 Assessments: • TJC and SJC: assessed on the same 2-point scale (0=absent; 1=present). • PtGADA: 100 mm VAS (0=very good, no symptoms; 100=very poor, severe symptoms). • CRP value calculated in mg/L. The 28 joints included the shoulders, elbows, wrists; metacarpophalangeal (MCP), thumb interphalangeal (IP), and proximal interphalangeal (PIP) joints of the hands; and the knees. Scores on the DAS28(CRP) range from 0 to approximately 10, where higher scores indicate more disease activity. Scores on the DAS28(CRP) range from 0 to approximately 10, where higher scores indicate more disease activity. A negative change in DAS28(CRP) score indicates an improvement in disease activity.
Time Frame: Baseline (Week 0 of Study RA0056) and Week 96 (Study RA0057)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 3 | 1 | 3 | 2 | 3 | 2 | 2 | 5
units on a scale | -3.2427 (1.74642) | -3.5767 | -2.5985 (2.16200) | -3.0999 (0.02877) | -1.7516 (2.03992) | -2.6451 (0.96108) | -3.3173 (3.23508) | -3.7982 (1.23889)

6. Secondary Outcome: The American College of Rheumatology (ACR) 20% (ACR20) Improvement Criteria Response Rate From Baseline (Week 0 of Study RA0056) to Week 12 of Study RA0057
Description: ACR20 represents at least 20% improvement from Baseline for each of TJC (68 joints) + SJC (66 joints) + at least 3 components of 5 for: PtGADA-VAS, Physician's Global Assessment of Disease Activity (PhGADA)-VAS, Patient's Assessment of Arthritis Pain (PAAP)-VAS, Health Assessment Questionnaire-Disability Index (HAQ-DI) and CRP. Assessments: • TJC and SJC: same 2-point scale (0=absent;1=present). • PtGADA: 100 mm VAS (0=very good, no symptoms;100=very poor, severe symptoms). • PhGADA: 100 mm VAS (0=very good, asymptomatic, no limitation of normal activities;100=very poor, very severe symptoms which were intolerable, inability to carry out all normal activities). • PAAP: 100 mm VAS (0=no pain;100=most severe pain). • HAQ-DI assessed degree of difficulty experienced in 8 domains of daily living activities (20 questions), its score (0-3) computed from item scores, with lower scores indicates less disability. • CRP in mg/L. Missing values were considered as non-responding status.
Time Frame: Baseline (Week 0 of Study RA0056) up to Week 12 (Study RA0057)
Population: FAS included all enrolled subjects who received at least 1 injection of CDP6038 (olokizumab) and in addition had at least 1 efficacy measurement in Study RA0057.
Measure: Number; unit: Percentage of responders
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 20 | 20 | 21 | 20 | 17 | 16 | 40 | 36
Percentage of responders | 40.0 | 50.0 | 76.2 | 35.0 | 58.8 | 50.0 | 47.5 | 52.8

7. Secondary Outcome: The ACR20 Improvement Criteria Response Rate From Baseline (Week 0 of Study RA0056) to Week 24 of Study RA0057
Description: ACR20 represents at least 20% improvement from Baseline for each of TJC (68 joints) + SJC (66 joints) + at least 3 components of 5 for: PtGADA-VAS, PhGADA-VAS, PAAP-VAS, HAQ-DI and CRP. Assessments: • TJC and SJC: same 2-point scale (0=absent;1=present). • PtGADA: 100 mm VAS (0=very good, no symptoms;100=very poor, severe symptoms). • PhGADA: 100 mm VAS (0=very good, asymptomatic, no limitation of normal activities;100=very poor, very severe symptoms which were intolerable, inability to carry out all normal activities). • PAAP: 100 mm VAS (0=no pain;100=most severe pain). • HAQ-DI assessed degree of difficulty experienced in 8 domains of daily living activities (20 questions), its score (0-3) computed from item scores, with lower scores indicates less disability. • CRP in mg/L. Missing values were considered as non-responding status.
Time Frame: Baseline (Week 0 of Study RA0056) up to Week 24 (Study RA0057)
Population: as for outcome 6
Measure: Number; unit: Percentage of responders
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 20 | 20 | 21 | 20 | 17 | 16 | 40 | 36
Percentage of responders | 40.0 | 50.0 | 66.7 | 30.0 | 47.1 | 62.5 | 42.5 | 63.9

8. Secondary Outcome: The ACR20 Improvement Criteria Response Rate From Baseline (Week 0 of Study RA0056) to Week 48 of Study RA0057
Description: as for outcome 7
Time Frame: Baseline (Week 0 of Study RA0056) up to Week 48 (Study RA0057)
Population: as for outcome 6
Measure: Number; unit: Percentage of responders
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 20 | 20 | 21 | 20 | 17 | 16 | 40 | 36
Percentage of responders | 40.0 | 30.0 | 42.9 | 35.0 | 47.1 | 43.8 | 25.0 | 50.0

9. Secondary Outcome: The ACR20 Improvement Criteria Response Rate From Baseline (Week 0 of Study RA0056) to Week 96 of Study RA0057
Description: as for outcome 7
Time Frame: Baseline (Week 0 of Study RA0056) up to Week 96 (Study RA0057)
Population: as for outcome 6
Measure: Number; unit: Percentage of responders
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 20 | 20 | 21 | 20 | 17 | 16 | 40 | 36
Percentage of responders | 15.0 | 5.0 | 9.5 | 5.0 | 11.8 | 12.5 | 2.5 | 13.9

10. Secondary Outcome: The ACR 50% (ACR50) Improvement Criteria Response Rate From Baseline (Week 0 of Study RA0056) to Week 12 of Study RA0057
Description: ACR50 represents at least 50% improvement from Baseline for each of TJC (68 joints) + SJC (66 joints) + at least 3 components of 5 for: PtGADA-VAS, PhGADA-VAS, PAAP-VAS, HAQ-DI and CRP. Assessments: • TJC and SJC: same 2-point scale (0=absent;1=present). • PtGADA: 100 mm VAS (0=very good, no symptoms;100=very poor, severe symptoms). • PhGADA: 100 mm VAS (0=very good, asymptomatic, no limitation of normal activities;100=very poor, very severe symptoms which were intolerable, inability to carry out all normal activities). • PAAP: 100 mm VAS (0=no pain;100=most severe pain). • HAQ-DI assessed degree of difficulty experienced in 8 domains of daily living activities (20 questions), its score (0-3) computed from item scores, with lower scores indicates less disability. • CRP in mg/L. Missing values were considered as non-responding status.
Time Frame: Baseline (Week 0 of Study RA0056) up to Week 12 (Study RA0057)
Population: as for outcome 6
Measure: Number; unit: Percentage of responders
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 20 | 20 | 21 | 20 | 17 | 16 | 40 | 36
Percentage of responders | 25.0 | 15.0 | 33.3 | 15.0 | 17.6 | 18.8 | 27.5 | 38.9

11. Secondary Outcome: The ACR50 Improvement Criteria Response Rate From Baseline (Week 0 of Study RA0056) to Week 24 of Study RA0057
Description: as for outcome 10
Time Frame: Baseline (Week 0 of Study RA0056) up to Week 24 (Study RA0057)
Population: as for outcome 6
Measure: Number; unit: Percentage of responders
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 20 | 20 | 21 | 20 | 17 | 16 | 40 | 36
Percentage of responders | 20.0 | 20.0 | 33.3 | 15.0 | 11.8 | 43.8 | 25.0 | 41.7

12. Secondary Outcome: The ACR50 Improvement Criteria Response Rate From Baseline (Week 0 of Study RA0056) to Week 48 of Study RA0057
Description: ACR50 represents at least 50% improvement from Baseline for each of TJC (68 joints) + SJC (66 joints) + at least 3 components of 5 for: PtGADA-VAS, PhGADA-VAS, PAAP-VAS, HAQ-DI and CRP. Assessments: • TJC and SJC: same 2-point scale (0=absent;1=present). • PtGADA: 100 mm VAS (0=very good, no symptoms;100=very poor, severe symptoms). • PhGADA: 100 mm VAS (0=very good, asymptomatic, no limitation of normal activities;100=very poor, very severe symptoms which were intolerable, inability to carry out all normal activities). • PAAP: 100 mm VAS (0=no pain;100=most severe pain). • HAQ-DI assessed degree of difficulty experienced in 8 domains of daily living activities (20 questions), its score (0-3) computed from item scores, with lower scores meaning less disability. • CRP in mg/L. Missing values were considered as non-responding status.
Time Frame: Baseline (Week 0 of Study RA0056) up to Week 48 (Study RA0057)
Population: as for outcome 6
Measure: Number; unit: Percentage of responders
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 20 | 20 | 21 | 20 | 17 | 16 | 40 | 36
Percentage of responders | 10.0 | 15.0 | 28.6 | 20.0 | 35.3 | 31.3 | 15.0 | 33.3

13. Secondary Outcome: The ACR50 Improvement Criteria Response Rate From Baseline (Week 0 of Study RA0056) to Week 96 of Study RA0057
Description: as for outcome 10
Time Frame: Baseline (Week 0 of Study RA0056) up to Week 96 (Study RA0057)
Population: as for outcome 6
Measure: Number; unit: Percentage of responders
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 20 | 20 | 21 | 20 | 17 | 16 | 40 | 36
Percentage of responders | 10.0 | 5.0 | 4.8 | 0.0 | 11.8 | 6.3 | 2.5 | 8.3

14. Secondary Outcome: The ACR 70% (ACR70) Improvement Criteria Response Rate From Baseline (Week 0 of Study RA0056) to Week 12 of Study RA0057
Description: ACR70 represents at least 70% improvement from Baseline for each of TJC (68 joints) + SJC (66 joints) + at least 3 components of 5 for: PtGADA-VAS, PhGADA-VAS, PAAP-VAS, HAQ-DI and CRP. Assessments: • TJC and SJC: same 2-point scale (0=absent;1=present). • PtGADA: 100 mm VAS (0=very good, no symptoms;100=very poor, severe symptoms). • PhGADA: 100 mm VAS (0=very good, asymptomatic, no limitation of normal activities;100=very poor, very severe symptoms which were intolerable, inability to carry out all normal activities). • PAAP: 100 mm VAS (0=no pain;100=most severe pain). • HAQ-DI assessed degree of difficulty experienced in 8 domains of daily living activities (20 questions), its score (0-3) computed from item scores, with lower scores indicates less disability. • CRP in mg/L. Missing values were considered as non-responding status.
Time Frame: Baseline (Week 0 of Study RA0056) up to Week 12 (Study RA0057)
Population: as for outcome 6
Measure: Number; unit: Percentage of responders
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 20 | 20 | 21 | 20 | 17 | 16 | 40 | 36
Percentage of responders | 10.0 | 5.0 | 19.0 | 5.0 | 0.0 | 18.8 | 15.0 | 13.9

15. Secondary Outcome: The ACR70 Improvement Criteria Response Rate From Baseline (Week 0 of Study RA0056) to Week 24 of Study RA0057
Description: as for outcome 14
Time Frame: Baseline (Week 0 of Study RA0056) up to Week 24 (Study RA0057)
Population: as for outcome 6
Measure: Number; unit: Percentage of responders
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 20 | 20 | 21 | 20 | 17 | 16 | 40 | 36
Percentage of responders | 10.0 | 15.0 | 19.0 | 5.0 | 0.0 | 12.5 | 10.0 | 25.0

16. Secondary Outcome: The ACR70 Improvement Criteria Response Rate From Baseline (Week 0 of Study RA0056) to Week 48 of Study RA0057
Description: as for outcome 14
Time Frame: Baseline (Week 0 of Study RA0056) up to Week 48 (Study RA0057)
Population: as for outcome 6
Measure: Number; unit: Percentage of responders
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 20 | 20 | 21 | 20 | 17 | 16 | 40 | 36
Percentage of responders | 5.0 | 5.0 | 23.8 | 10.0 | 11.8 | 6.3 | 10.0 | 13.9

17. Secondary Outcome: The ACR70 Improvement Criteria Response Rate From Baseline (Week 0 of Study RA0056) to Week 96 of Study RA0057
Description: as for outcome 14
Time Frame: Baseline (Week 0 of Study RA0056) up to Week 96 (Study RA0057)
Population: as for outcome 6
Measure: Number; unit: Percentage of responders
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 20 | 20 | 21 | 20 | 17 | 16 | 40 | 36
Percentage of responders | 5.0 | 0.0 | 4.8 | 0.0 | 5.9 | 0.0 | 2.5 | 5.6

18. Secondary Outcome: Percentage of Subjects With DAS28(CRP) <2.6 at Week 12 of Study RA0057
Description: DAS28(CRP) was calculated using the TJC and SJC from 28 joints, the PtGADA-VAS, and CRP according to the formula: DAS28(CRP)=0.56 * (TJC)^1/2 + 0.28 * (SJC)^1/2 + 0.36 * ln(CRP[mg/L]+1) + 0.014 * PtGADA + 0.96 Assessments: • TJC and SJC: assessed on the same 2-point scale (0=absent; 1=present). • PtGADA: 100 mm VAS (0=very good, no symptoms; 100=very poor, severe symptoms). • CRP value calculated in mg/L. The 28 joints included the shoulders, elbows, wrists; metacarpophalangeal (MCP), thumb interphalangeal (IP), and proximal interphalangeal (PIP) joints of the hands; and the knees. Scores on the DAS28(CRP) range from 0 to approximately 10, where higher scores indicate more disease activity. A DAS28(CRP) score less than 2.6 implies remission.
Time Frame: Week 12 (Study RA0057)
Population: as for outcome 6
Measure: Number; unit: Percentage of subjects
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 20 | 20 | 21 | 20 | 17 | 16 | 40 | 36
Percentage of subjects | 25.0 | 30.0 | 38.1 | 25.0 | 0 | 18.8 | 25.0 | 25.0

19. Secondary Outcome: Percentage of Subjects With DAS28(CRP) <2.6 at Week 24 of Study RA0057
Description: as for outcome 18
Time Frame: Week 24 (Study RA0057)
Population: as for outcome 6
Measure: Number; unit: Percentage of subjects
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 20 | 20 | 21 | 20 | 17 | 16 | 40 | 36
Percentage of subjects | 25.0 | 35.0 | 33.3 | 25.0 | 17.6 | 12.5 | 20.0 | 33.3

20. Secondary Outcome: Percentage of Subjects With DAS28(CRP) <2.6 at Week 48 of Study RA0057
Description: as for outcome 18
Time Frame: Week 48 (Study RA0057)
Population: as for outcome 6
Measure: Number; unit: Percentage of subjects
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 20 | 20 | 21 | 20 | 17 | 16 | 40 | 36
Percentage of subjects | 20.0 | 30.0 | 23.8 | 20.0 | 29.4 | 12.5 | 15.0 | 22.2

21. Secondary Outcome: Percentage of Subjects With DAS28(CRP) <2.6 at Week 96 of Study RA0057
Description: as for outcome 18
Time Frame: Week 96 (Study RA0057)
Population: as for outcome 6
Measure: Number; unit: Percentage of subjects
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 20 | 20 | 21 | 20 | 17 | 16 | 40 | 36
Percentage of subjects | 10.0 | 5.0 | 9.5 | 5.0 | 11.8 | 0 | 2.5 | 8.3

22. Secondary Outcome: Percentage of Subjects With DAS28(CRP) ≤3.2 at Week 12 of Study RA0057
Description: DAS28(CRP) was calculated using the TJC and SJC from 28 joints, the PtGADA-VAS, and CRP according to the formula: DAS28(CRP)=0.56 * (TJC)^1/2 + 0.28 * (SJC)^1/2 + 0.36 * ln(CRP[mg/L]+1) + 0.014 * PtGADA + 0.96 Assessments: • TJC and SJC: assessed on the same 2-point scale (0=absent; 1=present). • PtGADA: 100 mm VAS (0=very good, no symptoms; 100=very poor, severe symptoms). • CRP value calculated in mg/L. The 28 joints included the shoulders, elbows, wrists; metacarpophalangeal (MCP), thumb interphalangeal (IP), and proximal interphalangeal (PIP) joints of the hands; and the knees. Scores on the DAS28(CRP) range from 0 to approximately 10, where higher scores indicate more disease activity. A DAS28(CRP) score less than or equal to (<=) 3.2 implies low disease activity.
Time Frame: Week 12 (Study RA0057)
Population: as for outcome 6
Measure: Number; unit: Percentage of subjects
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 20 | 20 | 21 | 20 | 17 | 16 | 40 | 36
Percentage of subjects | 35.6 | 40.0 | 52.4 | 30.0 | 17.6 | 25.0 | 35.0 | 44.4

23. Secondary Outcome: Percentage of Subjects With DAS28(CRP) ≤3.2 at Week 24 of Study RA0057
Description: DAS28(CRP) was calculated using the TJC and SJC from 28 joints, the PtGADA-VAS, and CRP according to the formula: DAS28(CRP)=0.56 * (TJC)^1/2 + 0.28 * (SJC)^1/2 + 0.36 * ln(CRP[mg/L]+1) + 0.014 * PtGADA + 0.96 Assessments: • TJC and SJC: assessed on the same 2-point scale (0=absent; 1=present). • PtGADA: 100 mm VAS (0=very good, no symptoms; 100=very poor, severe symptoms). • CRP value calculated in mg/L. The 28 joints included the shoulders, elbows, wrists; metacarpophalangeal (MCP), thumb interphalangeal (IP), and proximal interphalangeal (PIP) joints of the hands; and the knees. Scores on the DAS28(CRP) range from 0 to approximately 10, where higher scores indicate more disease activity. A DAS28(CRP) score <=3.2 implies low disease activity.
Time Frame: Week 24 (Study RA0057)
Population: as for outcome 6
Measure: Number; unit: Percentage of subjects
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 20 | 20 | 21 | 20 | 17 | 16 | 40 | 36
Percentage of subjects | 35.0 | 40.0 | 38.1 | 30.0 | 23.5 | 37.5 | 35.0 | 50.0

24. Secondary Outcome: Percentage of Subjects With DAS28(CRP) ≤3.2 at Week 48 of Study RA0057
Description: as for outcome 23
Time Frame: Week 48 (Study RA0057)
Population: as for outcome 6
Measure: Number; unit: Percentage of subjects
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 20 | 20 | 21 | 20 | 17 | 16 | 40 | 36
Percentage of subjects | 25.0 | 45.0 | 23.8 | 25.0 | 29.4 | 18.8 | 22.5 | 47.2

25. Secondary Outcome: Percentage of Subjects With DAS28(CRP) ≤3.2 at Week 96 of Study RA0057
Description: as for outcome 23
Time Frame: Week 96 (Study RA0057)
Population: as for outcome 6
Measure: Number; unit: Percentage of subjects
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 20 | 20 | 21 | 20 | 17 | 16 | 40 | 36
Percentage of subjects | 15.0 | 5.0 | 9.5 | 5.0 | 11.8 | 0 | 2.5 | 11.1

26. Secondary Outcome: Change From Baseline (Week 0 of Study RA0056) in the Clinical Disease Activity Index (CDAI) to Week 48 of Study RA0057
Description: CDAI was calculated using the TJC (28 joints), SJC (28 joints), PtGADA-VAS and PhGADA-VAS, according to the following formula: SJC + TJC + PtGADA + PhGADA Assessments: • TJC and SJC: assessed on the same 2-point scale (0=absent; 1=present). • PtGADA: 10 cm VAS (0=very good, no symptoms; 100=very poor, severe symptoms). • PhGADA: 10 cm VAS (0=very good, asymptomatic and no limitation of normal activities; 100=very poor, very severe symptoms which were intolerable and inability to carry out all normal activities). The 28 joints included the shoulders, elbows, wrists; metacarpophalangeal (MCP), thumb interphalangeal (IP), and proximal interphalangeal (PIP) joints of the hands; and the knees. Total score range is from 0-100, with the high scores representing high disease activity. A negative change in CDAI score indicates an improvement in disease activity.
Time Frame: Baseline (Week 0 of Study RA0056) and Week 48 (Study RA0057)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 10 | 13 | 14 | 10 | 12 | 10 | 20 | 23
units on a scale | -80.1000 (53.28425) [lower limit 53.28425] | -65.3373 (63.72098) [lower limit 63.72098] | -94.3335 (61.48562) [lower limit 61.48562] | -80.8077 (57.91606) [lower limit 57.91606] | -79.9231 (30.09849) [lower limit 30.09849] | -84.8378 (33.77586) [lower limit 33.77586] | -74.3315 (53.99274) [lower limit 53.99274] | -83.4950 (42.48396) [lower limit 42.48396]

27. Secondary Outcome: Change From Baseline (Week 0 of Study RA0056) in the CDAI to Week 96 of Study RA0057
Description: as for outcome 26
Time Frame: Baseline (Week 0 of Study RA0056) and Week 96 (Study RA0057)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 3 | 1 | 3 | 2 | 3 | 2 | 2 | 5
units on a scale | -108.0000 (66.77574) | -118.0000 | -89.0000 (55.97321) | -74.3846 (4.78657) | -74.0000 (55.74944) | -90.5000 (13.43503) | -104.5000 (126.57211) | -107.4000 (51.52960)

28. Secondary Outcome: Change From Baseline (Week 0 of Study RA0056) in the Simplified Disease Activity Index (SDAI) to Week 48 of Study RA0057
Description: SDAI was calculated using the TJC (28 joints), SJC (28 joints), PtGADA-VAS, PhGADA-VAS and CRP (in milligrams per decilitre [mg/dL]), according to the following formula: SJC + TJC + PtGADA + PhGADA + CRP (mg/dL) Assessments: • TJC and SJC: assessed on the same 2-point scale (0=absent; 1=present). • PtGADA: 10 cm VAS (0=very good, no symptoms; 100=very poor, severe symptoms). • PhGADA: 10 cm VAS (0=very good, asymptomatic and no limitation of normal activities; 100=very poor, very severe symptoms which were intolerable and inability to carry out all normal activities). • CRP range was from 0 to 10 mg/dL. The 28 joints included the shoulders, elbows, wrists; metacarpophalangeal (MCP), thumb interphalangeal (IP), and proximal interphalangeal (PIP) joints of the hands; and the knees. The SDAI score ranges from 0 to 86, with higher scores representing worse disease. A negative change in SDAI score indicates an improvement in disease activity.
Time Frame: Baseline (Week 0 of Study RA0056) and Week 48 (Study RA0057)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 10 | 13 | 13 | 10 | 12 | 10 | 20 | 23
units on a scale | -92.1000 (62.22799) [lower limit 62.22799] | -75.8757 (74.37825) [lower limit 74.37825] | -104.6668 (80.47988) [lower limit 80.47988] | -92.4077 (55.42723) [lower limit 55.42723] | -87.7564 (28.41084) [lower limit 28.41084] | -112.5378 (52.99896) [lower limit 52.99896] | -87.5815 (59.26016) [lower limit 59.26016] | -107.4080 (60.17362) [lower limit 60.17362]

29. Secondary Outcome: Change From Baseline (Week 0 of Study RA0056) in the SDAI to Week 96 of Study RA0057
Description: as for outcome 28
Time Frame: Baseline (Week 0 of Study RA0056) and Week 96 (Study RA0057)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
Number analyzed (Participants) | 3 | 1 | 3 | 2 | 3 | 2 | 2 | 5
units on a scale | -111.0000 (68.78953) | -125.0000 | -90.3333 (56.04760) | -91.8846 (29.53531) | -75.3333 (56.09219) | -147.5000 (77.07464) | -128.0000 (147.07821) | -143.4000 (80.28574)

ADVERSE EVENTS:
Time Frame: From Baseline (Week 0 of Study RA0057) until 30 days after the last dose (maximum up to 780 days)
Description: Reported TEAEs included adverse events that started or worsened after the first dose of CDP6038 (olokizumab) in Study RA0057 and within 30 days after the last dose.
Groups:
- RA0056 CDP6038 (Olokizumab) 240 mg q2w: CDP6038 (olokizumab) 240 mg administered q2w sc in Study RA0056, followed by switch to CDP6038 (olokizumab) 120 mg q2w sc at start of Study RA0057 (Week 12 of RA0056).
Arm/Group | RA0056 CDP6038 (Olokizumab) 120 mg q2w | RA0056 CDP6038 (Olokizumab) 120 mg q4w | RA0056 CDP6038 (Olokizumab) 240 mg q2w | RA0056 CDP6038 (Olokizumab) 240 mg q4w | RA0056 CDP6038 (Olokizumab) 60 mg q2w | RA0056 CDP6038 (Olokizumab) 60 mg q4w | RA0056 Placebo | RA0056 Tocilizumab 8 mg/kg q4w
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/21 | 0/20 | 0/17 | 1/16 | 1/40 | 0/36
Serious Adverse Events (participants affected / at risk) | 3/20 | 6/20 | 6/21 | 7/20 | 5/17 | 3/16 | 14/40 | 4/36
Other Adverse Events (participants affected / at risk) | 16/20 | 20/20 | 18/21 | 17/20 | 15/17 | 15/16 | 36/40 | 35/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RA0056 CDP6038 (Olokizumab) 120 mg q2w (N=20) | RA0056 CDP6038 (Olokizumab) 120 mg q4w (N=20) | RA0056 CDP6038 (Olokizumab) 240 mg q2w (N=21) | RA0056 CDP6038 (Olokizumab) 240 mg q4w (N=20) | RA0056 CDP6038 (Olokizumab) 60 mg q2w (N=17) | RA0056 CDP6038 (Olokizumab) 60 mg q4w (N=16) | RA0056 Placebo (N=40) | RA0056 Tocilizumab 8 mg/kg q4w (N=36)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression suicidal (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic foot infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incision site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal fusion surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Unevaluable event (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RA0056 CDP6038 (Olokizumab) 120 mg q2w (N=20) | RA0056 CDP6038 (Olokizumab) 120 mg q4w (N=20) | RA0056 CDP6038 (Olokizumab) 240 mg q2w (N=21) | RA0056 CDP6038 (Olokizumab) 240 mg q4w (N=20) | RA0056 CDP6038 (Olokizumab) 60 mg q2w (N=17) | RA0056 CDP6038 (Olokizumab) 60 mg q4w (N=16) | RA0056 Placebo (N=40) | RA0056 Tocilizumab 8 mg/kg q4w (N=36)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (6) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Macrocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Monocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 7 (8) | 4 (4)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 3 (4) | 1 (5) | 0 (0) | 1 (1) | 5 (5) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 3 (4) | 1 (1) | 3 (3) | 5 (7) | 3 (4)
Cellulitis (Infections and infestations) | 1 (1) | 2 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Ear infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (3) | 6 (10) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 3 (5)
Oral herpes (Infections and infestations) | 1 (2) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Otitis media (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 4 (4) | 6 (7)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3) | 9 (12) | 2 (2) | 4 (6) | 3 (3) | 7 (10) | 5 (9)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (3) | 6 (24) | 2 (2) | 2 (3) | 3 (5) | 5 (12) | 5 (11)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (3)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vaginitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 1 (1) | 2 (3) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (4)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (5) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (5) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (5) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 2 (8)
Lipids increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 2 (2)
Low density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Mammogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Red cell distribution width increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (6) | 0 (0) | 2 (2) | 3 (5) | 3 (3) | 1 (2) | 5 (5) | 6 (10)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 2 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 3 (5)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3) | 1 (2) | 3 (3) | 1 (1) | 3 (3) | 3 (3) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 7 (7) | 4 (4)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendon calcification (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (5) | 6 (7) | 1 (2) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 4 (8)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
Pyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (6) | 3 (3) | 2 (2) | 1 (1) | 4 (6) | 6 (7) | 5 (8)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Laryngeal mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (5)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 3 (4) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 5 (5)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 2 (2)
Injection site reaction (General disorders) | 2 (2) | 2 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 6 (8) | 8 (14)
Oedema peripheral (General disorders) | 1 (2) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 2 (3)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (9) | 1 (2) | 2 (4) | 2 (2)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (11) | 1 (1) | 1 (16) | 3 (18) | 3 (21)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The clinical trial was terminated early as a result of a strategic UCB decision to out-license the study drug for further development. As a result, only small numbers of subjects were still in the study past the Week 48 time point.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. The Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.